CLINICAL TRIAL: NCT07407699
Title: Isulin Resistance as a Mediator of Chronic Pain in Postmenopausal Women: Effects of a Combined Exercise Program on Metabolic and Inflammatory Mechanisms
Brief Title: Exercise, Insulin Resistance, and Chronic Pain in Postmenopausal Women.
Acronym: EX-PAIN-MENO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Gabriela Carrion Caldeira Ribeiro, Masters, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOUTORADO_FCT_UNESP_2026
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Postmenopausal; Insulin Resistance
MeSH Terms: conditions — Chronic Pain; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Postmenopausal women undergoing a supervised combined exercise program (aerobic, resistance, and mind-body exercise).
  Interventions: Behavioral: Combined Exercise Program; Other: Usual Care Group
- Control Group (No Intervention): Postmenopausal women who will continue receiving usual care without participation in a structured exercise program during the study period.

INTERVENTIONS:
Behavioral: Combined Exercise Program — Participants allocated to the intervention group will take part in a supervised combined exercise program, performed twice weekly for 12 months. Each session will last approximately 60 minutes and will include aerobic exercise, resistance training, and mind-body exercise.
  Aerobic training will consist of walking or cycling at moderate intensity, monitored by heart rate. Resistance training will involve multi-joint exercises using body weight and elastic bands, with progressive overload. Mind-body exercise will be performed using restorative yoga techniques. Exercise sessions will be supervised by a trained physiotherapist.
  Arms: Intervention group
Other: Usual Care Group — Participants allocated to the control group will continue with their usual care and daily activities, without participation in any structured or supervised exercise program during the study period.
  Arms: Intervention group

SUMMARY:
This study aims to investigate the effects of a combined exercise program on chronic pain in postmenopausal women, considering insulin resistance as a potential physiological mediator. The intervention will assess changes in pain intensity, metabolic and inflammatory biomarkers, psychosocial factors, and body composition. The findings may contribute to understanding the metabolic mechanisms underlying chronic pain in postmenopausal women and support exercise as a non-pharmacological therapeutic strategy.

DETAILED DESCRIPTION:
Postmenopausal women experience a high prevalence of chronic musculoskeletal pain, potentially influenced by hormonal depletion, metabolic dysfunction, and low-grade systemic inflammation. Insulin resistance has been associated with inflammatory processes and may contribute to peripheral and central sensitization mechanisms involved in chronic pain.

This randomized controlled trial will evaluate the effects of a combined exercise intervention, including aerobic, resistance, and mind-body components, on pain intensity and related outcomes in postmenopausal women with chronic pain. Secondary outcomes include metabolic markers, inflammatory biomarkers, psychosocial variables, and body composition. Insulin resistance will be explored as a mediator of pain modulation following the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, defined as between 12 months and 5 years since the last menstrual period.
* Not using hormone replacement therapy.
* Not engaged in regular physical exercise (defined as more than once per week in the last months).
* With or without insulin resistance.

Exclusion Criteria:

* Diagnosis of neurological diseases (e.g., Parkinson's disease, multiple sclerosis, or stroke sequelae).
* Severe psychiatric disorders.
* Inflammatory autoimmune diseases (e.g., rheumatoid arthritis or systemic lupus erythematosus).
* Active neoplasms.
* Use of systemic corticosteroids or immunosuppressive drugs within the last three months.
* Severe decompensated cardiovascular disease.
* Any medical condition that contraindicates participation in physical exercise.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline and at 12 months following intervention
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), ranging from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Insulin Resistance assessed by Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline (pre-intervention) and after 12 months of intervention
  Insulin resistance will be evaluated using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), calculated from fasting glucose and fasting insulin levels.
Anxiety assessed by Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A) | Baseline and after 12 months of intervention
  Anxiety symptoms will be assessed using the Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A), ranging from 0 to 21, with higher scores indicating greater anxiety symptoms.
Depression assessed by Hospital Anxiety and Depression Scale - Depression subscale (HADS-D) | Baseline and after 12 months of intervention
  Depressive symptoms will be assessed using the Hospital Anxiety and Depression Scale - Depression subscale (HADS-D), ranging from 0 to 21, with higher scores indicating greater depressive symptoms.
Pain catastrophizing assessed by Pain Catastrophizing Scale (PCS) | Baseline and after 12 months of intervention
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS), ranging from 0 to 52, with higher scores indicating greater catastrophizing.
Pain self-efficacy assessed by Pain Self-Efficacy Questionnaire (PSEQ) | Baseline and after 12 months of intervention
  Self-efficacy related to pain management will be assessed using the Pain Self-Efficacy Questionnaire (PSEQ), ranging from 0 to 60, with higher scores indicating greater self-efficacy.
Quality of life assessed by Short Form Health Survey (SF-36) | Baseline and after 12 months of intervention
  Quality of life will be assessed using the Short Form Health Survey (SF-36), with scores ranging from 0 to 100, where higher scores indicate better health-related quality of life.
Sleep quality assessed by Pittsburgh Sleep Quality Index (PSQI) | Baseline and after 12 months of intervention
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), ranging from 0 to 21, with higher scores indicating worse sleep quality.
Body weight | Baseline and after 12 months of intervention
  Body weight will be measured using a calibrated scale and expressed in kilograms (kg).
Body fat percentage assessed by dual-energy X-ray absorptiometry (DEXA) | Baseline and after 12 months of intervention
  Body fat percentage will be assessed using dual-energy X-ray absorptiometry (DEXA). Values will be expressed as percentage (%), with higher values indicating greater body fat.
Total fat mass assessed by dual-energy X-ray absorptiometry (DEXA) | Baseline and after 12 months of intervention
  Total fat mass will be assessed using dual-energy X-ray absorptiometry (DEXA) and expressed in kilograms (kg).
Total lean mass assessed by dual-energy X-ray absorptiometry (DEXA) | Baseline and after 12 months of intervention
  Total lean mass will be assessed using dual-energy X-ray absorptiometry (DEXA) and expressed in kilograms (kg). Higher values indicate greater lean mass.